CLINICAL TRIAL: NCT06770842
Title: Safety and Efficacy of Ropeginterferon Alfa-2b in Combination With Ruxolitinib in Patients With Myelofibrosis Demonstrating Suboptimal Response to Ruxolitinib Monotherapy
Brief Title: Ropeginterferon Alfa 2b Plus Ruxolitinib for Myelofibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1101RUXMF
Record Dates: First submitted 2024-12-20; First posted 2025-01-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-12

CONDITIONS: Primary Myelofibrosis (PMF); Post Polycythemia Myelofibrosis (PPV MF); Post Essential Thrombocythaemia Myelofibrosis (PET-MF)
Keywords: Ruxolitinib; Ropeginterferon alfa 2b; Myelofibrosis; Ruxolitinib failiure
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ropeginterferon alfa 2b (Experimental): Ropeginterferon alfa 2b is administered subcutaneously once every 2 weeks in addition to standard of care with Ruxolitinib which will be self-administered orally as described below. Both medications will continue uninterrupted in 28-day cycles. Subjects will continue combination treatment through the Initial Treatment Period (ITP) (first 6 cycles), which includes a Qualification Assessment. Those deriving clinical benefit in the opinion of the treating physician may continue receiving combination treatment in the Additional Treatment Period (6 cycles). Qualification Assessments will be performed at the end of each Additional Treatment Period, which is iterative, and may repeat for as long as clinical benefit is sustained, at the discretion of the treating physician.
  Interventions: Drug: Ropeginterferon alfa-2b (BESREMi®)

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b (BESREMi®) — Ropeginterferon alfa 2b is administered subcutaneously once every 2 weeks. The dosing will be 250mcg at Week 0, 350mcg at Week 2, 500mcg at Week 4, and 500mcg every 2 weeks thereafter

SUMMARY:
In this open-label single arm phase 2 study, approximately 20 patients with MF demonstrating suboptimal response to ruxolitinib monotherapy will be enrolled. Patients will continue to receive ruxolitinib at a stable dose and ropeginterferon alfa 2b will be added to the regimen.

DETAILED DESCRIPTION:
Ropeginterferon alfa 2b is administered subcutaneously once every 2 weeks. Ruxolitinib is self-administered orally as part of standard of care. BSubjects will continue combination treatment through the Initial Treatment Period (ITP) (first 6 cycles), which includes a Qualification Assessment. Those deriving clinical benefit in the opinion of the treating physician may continue receiving combination treatment in the Additional Treatment Period (6 cycles). Qualification Assessments will be performed at the end of each Additional Treatment Period, which is iterative, and may repeat for as long as clinical benefit is sustained, at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Age ≥18 years
* Diagnosis of Overt Myelofibrosis (primary, post-ET, or post-PV) per World Health Organization (WHO) 2022 diagnostic criteria
* Intermediate-1, Intermediate-2, or high-risk disease by Dynamic International Prognostic Scoring System (DIPSS)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Platelet count ≥75 x 109/L prior to dosing on Cycle 1 Day 1
* Absolute neutrophil count ≥0.5 x 109/L prior to dosing on Cycle 1 Day 1
* Peripheral blast count ≤10% prior to dosing on Cycle 1 Day 1
* Women of childbearing potential and fertile men must agree to use an approved method of contraception from screening until 30 days after the last dose of ropeginterferon and ruxolitinib.
* Patients with suboptimal response to ruxolitinib as per one of the below:

  i. Relapsed: Ruxolitinib treatment for ≥3 months with spleen regrowth, defined as <10% SVR or <30% decrease in spleen size from baseline, following an initial response* ii. Refractory: Ruxolitinib treatment for ≥3 months with <10% SVR or <30% decrease in spleen size from baseline.

  * Response to ruxolitinib is defined as a ≥35% reduction in spleen volume from baseline, or a ≥50% reduction in spleen size for baseline spleen sizes >10 cm below left costal margin (LCM); a non-palpable spleen for baseline spleen sizes between 5-10 cm below LCM; or not eligible for spleen response for baseline spleen <5 cm below LCM.

Exclusion Criteria:

Subjects will not be eligible for participation if they meet any of the following exclusion criteria:

* Prior or current use of interferon alfa (IFNα) preparations for MPN
* Patients currently on other investigational therapy (ies)
* Contraindications or hypersensitivity to IFNα preparations
* History of organ and haematopoietic stem cell transplantation
* History of splenectomy
* Pregnant or lactating females, or females planning to become pregnant at any time during the study
* Documented autoimmune disease at screening
* Infection with human immunodeficiency virus (HIV)
* Active and uncontrolled infections with hepatitis B virus (HBV) and hepatitis C virus (HCV). Please note that patients on antiviral therapy with undetectable HBV DNA and HCV RNA may be recruited.
* Evidence of severe retinopathy including but not limited to macular degeneration, diabetic retinopathy and hypertensive retinopathy.
* History of clinically significant neuropsychiatric conditions including but not limited to depression and epilepsy.
* Clinically significant neuropsychiatric conditions including but not limited to depression and epilepsy.
* Concurrent second active and non-stable malignancy (patients with a concurrent second active but stable malignancy, i.e., non-melanoma skin cancers, are eligible)
* Evidence of alcohol or drug abuse within 6 months
* Evidence at the time of Screening of significant renal or hepatic insufficiency (unless due to hemolysis) as defined by any of the following local lab parameters:

  * Calculated glomerular filtration rate (GFR; using the Cockcroft-Gault equation) <40 mL/min or serum creatinine >1.5 x the local upper limit of normal
  * Aspartate transaminase (AST) or alanine aminotransferase (ALT) ≥2.5 x the local upper limit of normal
* Unwilling or unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 24 months
  Enumeration and description of adverse events (AEs), including determination of dose limiting toxicities (DLTs), serious adverse events (SAEs), and other AEs

SECONDARY OUTCOMES:
Spleen volume change at 24 weeks | 24 weeks
  Proportion of patients who experience a spleen length reduction by palpation of ≥30% OR spleen volume reduction (SVR) of ≥35% by MRI or CT by 24 weeks of treatment
Symptom response at 24 weeks | 24 weeks
  Proportion of patients who describe a ≥50% reduction in symptom burden by the myelofibrosis symptom assessment form (MFSAF) by 24 weeks of treatment. The MFSAF has a scale of 0-70 where a higher score indicates worse outcome.

OTHER OUTCOMES:
Rate of molecular responses | 24 months
  Changes in allelic burden of JAK2V617F, MPL, CALR or other driver mutations will be assessed. A molecular responses is assessed using the International Working Group of Myeloproliferative Neoplasm Research and Treatment Criteria.
Rate of morphologic response | 24 months
  Changes in bone marrow morphology (cellularity, erythroid, myeloid, megakaryocyte, reticulin and fibrosis) during treatment. Response is assessed using the International Working Group of Myeloproliferative Neoplasm Research and Treatment Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Gill, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No